CLINICAL TRIAL: NCT00819598
Title: Pilot Study to Determine the Optimal Oscillometric-Based Technique for Measurement of Ankle Blood Pressures for the Ankle-brachial Index
Brief Title: Pilot Study to Determine the Optimal Technique for Measurement of Ankle Blood Pressures
Status: Completed | Type: Observational
Sponsor: Summit Doppler Systems, Inc. (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Dr. Heather Gornik, Cleveland Clinic
Other Study IDs: CCF IRB 08-823
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SUSPECTED ARTERIAL DISEASE
  Interventions: Procedure: BLOOD PRESSURE MEASURMENT; Procedure: BLOOD PRESSURE MEASUREMENT

INTERVENTIONS:
Procedure: BLOOD PRESSURE MEASURMENT — Blood pressures using Doppler and oscillometric methods will be obtained at each limb and on one toe from each foot.
Procedure: BLOOD PRESSURE MEASUREMENT — Blood pressure measurements will be taken at each limb (arm and ankle) with Doppler and oscillometric based methods.

SUMMARY:
Peripheral arterial disease (PAD) is a highly prevalent medical condition. Patients with PAD are usually diagnosed on the basis of the ankle-brachial index. The ankle-brachial index is the ratio of ankle pressure to arm pressure based on measurement of blood pressures in the arms and legs using a Doppler device. The need for dedicated equipment and trained personnel, along with the time required to perform the test, have been identified as barriers to widespread implementation of ankle-brachial index screening. The use of automated oscillometric devices for blood pressure measurement and determination of the ankle-brachial index has been applied with variable success. It will be beneficial to investigate a reliable oscillometric-based procedure that can accurately measure leg pressures for the ankle-brachial index across the entire spectrum of PAD severity.

The purpose of this study is to determine the optimal oscillometric-based technique for estimation of Doppler-derived systolic arm and ankle blood pressures for calculation of the ankle-brachial index in patients with and without PAD.

Subjects with suspected arterial disease in the non-invasive lab will be enrolled. Arm, ankle, and toe pressure measurements will be made in the supine position using Doppler, oscillometric methods, and photoplethysmographic sensor. Arm and ankle pressures from a subset of subjects will be obtained in both seated and supine positions. The ankle-brachial index and toe-brachial index will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 50 years of age
* Ambulatory outpatient
* Referred to non-invasive Vascular Laboratory for evaluation of suspected arterial disease.

Exclusion Criteria:

* Unable to give informed consent
* Unable to lie supine for at least 15 minutes

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to Cleveland Clinic's non-invasive vascular lab
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather L Gornik, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States